CLINICAL TRIAL: NCT04499131
Title: Exploratory Study on the Impact of Different Doses and Route of Administration of Exogenous Progesterone in Artificial Endometrial Preparation Cycles on Endometrial Structure and Function
Brief Title: Impact of Different Doses and Routes of Exogenous Progesterone Administration on Endometrial Receptivity Parameters
Acronym: PROGENDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1901-VLC-014-EL
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female; ENDOMETRIAL RECEPTIVITY
Keywords: Luteal phase; Artificial endometrial preparation cycle; Progesterone; Endometrial gene expression; Endometrial receptivity
MeSH Terms: conditions — Infertility, Female | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Exploratory, unicentric, with blind evaluators, randomized to six parallel arms in ratio 1:1:1:1:1:1 clinical trial conducted in healthy volunteers under an artificial endometrial preparation cycle and luteal phase support with exogenous progesterone administered by different doses and routes or natural menstrual cycles.
Who Masked: Investigator
Masking Description: Patients will be evaluated by blinded gynecologist in order to prevent the application of personal criteria and protect the consistence of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- I: Artificial endometrial preparation cycle (Experimental): Artificial endometrial preparation cycle with estrogens and vaginal natural micronized progesterone 400mg/12h
  Interventions: Drug: Progesterone
- II: Artificial endometrial preparation cycle (Experimental): Artificial endometrial preparation cycle with estrogens and subcutaneous natural progesterone 25mg/24h
  Interventions: Drug: Progesterone
- III: Artificial endometrial preparation cycle (Experimental): Artificial endometrial preparation cycle with estrogens and subcutaneous natural progesterone 25mg/12h
  Interventions: Drug: Progesterone
- IV: Artificial endometrial preparation cycle (Experimental): Artificial endometrial preparation cycle with estrogens and a combination of subcutaneous natural progesterone 25mg/24h + vaginal natural micronized progesterone 400mg/24h
  Interventions: Drug: Progesterone
- V: Artificial endometrial preparation cycle (Experimental): Artificial endometrial preparation cycle with estrogens and intramuscular natural progesterone 50mg/24h
  Interventions: Drug: Progesterone
- Natural menstrual cycle (Active Comparator): Natural menstrual cycle (without any exogenous steroid hormone Treatment)
  Interventions: Other: Artificial Cycle (no intervention)

INTERVENTIONS:
Drug: Progesterone — Subjects will undergo an artificial cycle with hormone replacement therapy (HRT) with the aim of comparing the endometrial gene expression profile in the different types of exogenous progesterone with different doses and routes of administration.
  Arms: I: Artificial endometrial preparation cycle; II: Artificial endometrial preparation cycle; III: Artificial endometrial preparation cycle; IV: Artificial endometrial preparation cycle; V: Artificial endometrial preparation cycle
Other: Artificial Cycle (no intervention) — Control group of 19 subjects in the context of a natural cycle with only endogenous progesterone present
  Arms: Natural menstrual cycle

SUMMARY:
After so many years conducting artificial endometrial preparation cycles for embryo transfer, there is no clear indication about which is the optimal dose of exogenous progesterone in this scenario to optimize the outcome. Taking into account that the luteal phase can be controlled by measuring serum P levels (not done until now), the next step is to find out which is the best dose and route of administration of exogenous progesterone for luteal phase in artificial cycles.

Therefore, the aim of this experimental study is to compare the endometrial function and structure, as well as the serum P levels according to the use of different types of exogenous progesterone available on the market depending on their doses and route of administration (vaginal, subcutaneous or intramuscular). The endometrial receptivity status will be compared in the different artificial cycles with the one observed in a natural cycle, without exogenous progesterone (only the endogenous one) as a control group.

Endometrial receptivity will be analysed by means of endometrial function and structure, but not by pregnancy outcome as in this study an embryo cannot be replaced in the uterus because an endometrial biopsy needs to be done to do this type of research.

ELIGIBILITY:
Inclusion Criteria

All women with no history of infertility who agree to participate in the study:

1. Age: 18-35 years old, both inclusive
2. Regular menstrual cycles
3. In good health and not suffering from any mental or medical condition(s) that would preclude participation in the study.

Exclusion Criteria

Subjects who meet one or more of the following will not be considered eligible to participate in the pilot study:

1. Simultaneous participation in other clinical studies that, at the researcher's criteria, could interfere with the results of this study.
2. Taking oral contraceptives in the three months prior to signing informed consent.
3. Presence of uterine pathology (submucosal or intramural myomas >4 cm deforming cavity, endometrial polyps or müllerian anomalies) or adnexal pathology (communicating hydrosalpinx).
4. Background of thrombosis, breast cancer, systemic diseases.
5. Those unable to comprehend the investigational nature of the proposed study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Endometrial gene expression profile | 12 months
  Determination of gene expression

SECONDARY OUTCOMES:
Histological dating of endometrial biopsies | 12 months
  Endometrial classification using Noyes criteria
Progesterone concentration in the endometrium | 12 months
  Endometrial progesterone values
Serum Progesterone concentrations | 12 months
  Blood serum progesterone values
Correlation between progesterone levels in blood and uterus. | 12 months
  Presence or Absence of correlation
Correlation between serum and uterine levels with endometrial transcriptome and histological dating | 12 months
  Presence or Absence of correlation

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Valenciano de Infertilidad Spain, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided